CLINICAL TRIAL: NCT01014130
Title: A Randomised Phase III Trial of Highly Conformal Hypofractionated Image Guided ("Stereotactic") Radiotherapy (HypoRT) Versus Conventionally Fractionated Radiotherapy (ConRT) for Inoperable Early Stage I Non-small Cell Lung Cancer (CHISEL)
Brief Title: Hypofractionated Radiotherapy (Stereotactic) Versus Conventional Radiotherapy for Inoperable Early Stage I Non-small Cell Lung Cancer (NSCLC)
Acronym: CHISEL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TROG 09.02
Record Dates: First submitted 2009-10-08; First posted 2009-11-16 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer; Hypofractionated; Stereotactic Radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 2 (Active Comparator): Conventionally Fractionated Radiotherapy (ConRT) - Standard of Care
  Interventions: Radiation: Conventionally Fractionated Radiotherapy (ConRT)
- Arm 1 (Experimental): Hypofractionated radiotherapy (HypoRT) - Investigational
  Interventions: Radiation: Hypofractionated radiotherapy (HypoRT)

INTERVENTIONS:
Radiation: Hypofractionated radiotherapy (HypoRT) — Highly conformal hypofractionated radiotherapy to a total dose of 54 Gy given in 3 fractions of 18 Gy each, delivered weekly on days 0, 7 and 14 with a maximum deviation of +/- 2 days from the specified time allowed.
  Other Names: HypoRT; Radiotherapy; RT
  Arms: Arm 1
Radiation: Conventionally Fractionated Radiotherapy (ConRT) — Standard radiotherapy to a total dose of 60-66 Gy prescribed to an isodose covering the PTV. It will be delivered as 30-33 fractions over a period of six to six and a half weeks. If the use of chemotherapy is the institutional practice for this group of patients, concurrent carboplatin and paclitaxel will be given weekly (paclitaxel (45mg/m2/wk) and carboplatin (AUC=2/wk) for 6 weeks.
  Other Names: ConRT; Radiotherapy; RT
  Arms: Arm 2

SUMMARY:
The purpose of this study is to investigate whether radiotherapy given as three large doses over a period of two weeks (hypofractionated radiotherapy) is more effective than standard radiotherapy for patients with non-small cell lung cancer that has not spread beyond the lung. Although surgery is the most effective treatment for early lung cancer, many patients are not fit enough for an operation. The alternative treatment to surgery is standard radiotherapy which is normally 'fractionated' that is, given as a number of small doses over a period of weeks. Experience has shown that many small treatments are safer than using a few large doses (hypofractionation) because there is less risk of damage to normal tissues.

Recent advances in technology have however resulted in greater accuracy and with it a reduction in the amount of normal tissue affected by the radiation, so the risks of hypo-fractionation damaging normal tissue are of less concern. Initial results obtained with hypo-fractionated radiotherapy for early stage non-small cell lung cancer indicate that it may be more effective in controlling the cancer. However, it has never been compared directly with standard fractionation in a randomised trial, so this study aims to determine if hypo-fractionation is more effective, results in longer life expectancy and if it is just as safe as standard fractionation.

DETAILED DESCRIPTION:
This is a multicentre randomised phase III trial comparing hypo-fractionated ("stereotactic') radiotherapy with conventional radiotherapy with or without chemotherapy in patients with inoperable stage 1 peripherally located non-small cell lung cancer.

The accepted standard of care for stage 1 non-small cell lung cancer (NSCLC), that is, T1 or T2 tumors that have not metastasised to the regional lymph nodes, is surgical resection. However, many patients with lung cancer have significant cardiovascular and respiratory co morbidities which render them unfit for an operation. For these patients, the standard of care is radiotherapy - conventional fractionation (ConRT) which is administered as 20-30 fractions over a period of four to six weeks. This reduces the likelihood of long term damage to incidentally irradiated normal tissues compared with non-fractionated treatment. Local failure for this method, varies considerably between reports ranging from 6-70% with a median value of 40% using a current best practice for inoperable NSCLC dose of about 60 Gy. Concomitant chemotherapy in addition to CF improves local progression free survival by 16% at two years compared with radiotherapy alone.

Highly conformal hypo-fractionated image guided radiotherapy is an emerging technically complex method for precision irradiation of stage 1 NSCLC using doses with a higher biological effect than can be achieved with standard treatment techniques. Although rates of local control using hypo-fractionation appear greater, there are risks with serious late toxicity. However, there is recent evidence that 54-57Gy delivered in 3 fractions can be delivered safely with no excessive toxicity, provided the tumour has a peripheral location, the chest wall is not included in the high dose volume and the treatment plan is highly conformal. Although hypo-fractionation under the above conditions appears to be tolerable, and is associated with high levels of local control, the results of a small number of phase II trials cannot be regarded as sufficient evidence to recommend it as the standard of care for inoperable stage I NSCLC.

This randomised phase III trial tests whether highly conformal hypo-fractionated image guided radiotherapy for peripherally located inoperable T1 and T2a NSCLC using a dose of 54 Gy in three fractions results in superior control of disease at the primary site compared with standard care consisting of conventionally fractionated radiotherapy with or without concomitant chemotherapy.

Treatment summary: Investigational arm - radical radiotherapy to a total dose of 54 Gy in 3 fractions of 18 Gy each, delivered weekly on days 0, 7 and 14 with a maximum deviation of +/- 2 days from the specified time allowed. Conventional arm - radical radiotherapy to a total dose of 60-66 Gy in 30-33 daily 2 Gy fractions over 6 weeks, with or without chemotherapy consisting of weekly carboplatin at an AUC of 2 and paclitaxel 45 mg/m2.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer diagnosed within 6 weeks prior to randomisation. The following primary cancer types are eligible: squamous cell carcinoma, adenocarcinoma, large cell carcinoma, bronchioloalveolar cell carcinoma, large cell neuroendocrine, and non-small cell carcinoma not otherwise specified.
* Aged 18 years or older.
* Disease stage T1N0 or T2aN0 (UICC TNM stage, 7th Ed, 2009), based on FDG PET/CT performed within 4-6 weeks prior to randomisation. T stage should be based on tumour size alone (i.e. no atelectasis).
* An ECOG performance status score of 0 or 1.
* The tumour has a peripheral location, defined as at least 1 cm beyond the mediastinum and 2 cm beyond the bifurcation of the lobar bronchi.
* Tumour is assessed as inoperable either i) because of unfitness for surgery as determined by the lung multidisciplinary team including thoracic surgeons and respiratory physicians or ii) because the patient refuses surgery.
* Female patients of childbearing potential and male patients must agree to use adequate contraception throughout the treatment phase of the study.
* If female and of childbearing potential, a negative pregnancy test was performed within 7 days prior to randomisation.
* Patient is expected to survive and be available for follow up for two years.
* Patient has provided written informed consent for participation in this trial prior to any protocol-specified procedures.
* Patient undergoing chemoradiation has satisfactory haematological and biochemical parameters as described below:

  * ANC ≥ 1.5 x 109,
  * Platelets ≥ 100 x 109/L, Hb ≥ 100g/L,
  * Creatinine clearance ≥ 40mls/min (patients with calculated creatinine clearance ≥ 40mls/min and < 60mls/min must have this confirmed by nuclear medicine GFR scan),
  * Bilirubin < 1.5 x ULN, and
  * ALT or AST < 2x ULN.

Exclusion Criteria:

* Centrally located tumours (< 1.0 cm from mediastinum or < 2.0 cm from bifurcation of lobar bronchus).
* Tumours within 1.0 cm of the chest wall.
* Prior chemotherapy.
* Previous radiotherapy to the area to be treated.
* Women who are pregnant or lactating.
* Patient with multiple synchronous primary tumours requiring radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Time to Local Failure | Completion of the two year follow up period for all patients.

SECONDARY OUTCOMES:
Overall Survival | Completion of the two year follow up period for all patients.
Cancer Specific survival | Completion of the two year follow up period for all patients.
Treatment Related Toxicity | Completion of the two year follow up period for all patients.
Quality of Life | Completion of the two year follow up period for all patients.

CONTACTS AND LOCATIONS:
Overall Officials: David Ball, MBBSMDRANZCR, Study Chair — Peter MacCallum Cancer Centre, Australia
Locations (19):
- Australia (16):
  - Canberra Hospital, Canberra, Australian Capital Territory
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Calvary Mater Hosipital, Newcastle, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Peter Maccallum Cancer Centre, Bendigo, Victoria
  - Austin Hospital, Heidelburg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Peter MacCallum Cancer Centre - Box Hill, Melbourne, Victoria
  - Peter MacCallum Cancer Centre - Morrabbin, Melbourne, Victoria
  - Alfred Hospital, Prahran, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- New Zealand (3):
  - Auckland Hospital, Epsom, Auckland
  - Midcentral District Health Board, Roslyn, Palmerston North
  - Canterbury District Health Board, Christchurch

REFERENCES:
- [Derived] Ball D, Mai GT, Vinod S, Babington S, Ruben J, Kron T, Chesson B, Herschtal A, Vanevski M, Rezo A, Elder C, Skala M, Wirth A, Wheeler G, Lim A, Shaw M, Schofield P, Irving L, Solomon B; TROG 09.02 CHISEL investigators. Stereotactic ablative radiotherapy versus standard radiotherapy in stage 1 non-small-cell lung cancer (TROG 09.02 CHISEL): a phase 3, open-label, randomised controlled trial. Lancet Oncol. 2019 Apr;20(4):494-503. doi: 10.1016/S1470-2045(18)30896-9. Epub 2019 Feb 12. PMID 30770291
- See also: Click here for more information about this study on the TROG website — http://www.trog.com.au